CLINICAL TRIAL: NCT01790139
Title: Oral Iohexol for Fecal/Fluid Tagging for CT Colonography: A Study to Improve Image Quality by Preventing Colonic Bubbles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Seong Ho Park, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2012-0584
Record Dates: First submitted 2013-02-07; First posted 2013-02-13 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Simethicone; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control group undergoes CT colonography after usual cathartic bowel cleansing using Colonlyte and fecal/fluid tagging. The tagging is done by administering orally 50 mL of iohexol (Omnipaque 350, GE Healthcare) 10 minutes after the completion of Colonlyte.
- Intervention-Oral Simethicone (Experimental): Intervention group undergoes CT colonography after usual cathartic bowel cleansing using Colonlyte, fecal/fluid tagging, and oral administration of simethicone. The tagging is done by administering orally 50 mL of iohexol (Omnipaque 350, GE Healthcare) 10 minutes after the completion of Colonlyte. As the interventional procedure in this intervention group, 10 mL of simethicone is administered orally immediately following the administration of iohexol.
  Interventions: Drug: Oral simethicone

INTERVENTIONS:
Drug: Oral simethicone — 10 mL of simethicone is administered as an agent to prevent colonic bubbles
  Other Names: Simethicone manufactured by Taejoon Pharm Co., Ltd.
  Arms: Intervention-Oral Simethicone

SUMMARY:
To determine whether colonic bubbles associated with CT colonography performed with iohexol for fecal/fluid tagging could be reduced by adding simethicone to the standard cathartic preparation.

DETAILED DESCRIPTION:
CT colonography (CTC) is a recently developed radiological examination to find colorectal neoplasia. Fecal/fluid tagging using oral administration of contrast is an essential procedure for CTC. Iohexol, which has recently started being used as an agent for fecal/fluid tagging, has great advantages as it has much more tolerable taste and much lower rates of adverse effects such as clamping or diarrhea compared with traditionally used Gastrografin/Gastroview. However, iohexol is frequently associated with an occurrence of a lot of bubbles in the colon, which makes CTC interpretation more time-consuming and laborious.

Past experience in colonoscopy field suggests that simethicone, a safety-proven highly inexpensive over-the-counter medicine, might resolve this issue. Given the fact that patient convenience is an important factor for a successful CTC and the fact that time-intensive nature of CTC interpretation is one of the major deterrents to wide spread adoption of CTC while CTC also needs to be as time efficient as possible in order to effectively serve the role of population screening for colorectal cancer, investigating the effect of simethicone to prevent the colonic bubbles on the time efficiency of CTC interpretation would be important. If simethicone can resolve the colonic bubble problem, CTC can be performed more conveniently for the patients as well as for the interpreting radiologists.

This study is to determine whether colonic bubbles associated with CT colonography performed with iohexol for fecal/fluid tagging could be reduced by adding simethicone to the standard cathartic preparation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are schedule to undergo colonoscopy for a suspicion of colonic neoplasia at the investigators' institution
* Those who agree to participate in the study

Exclusion Criteria:

* Colonoscopy for reasons other than detecting colonic neoplasia, e.g. evaluation of inflammatory bowel disease
* Contraindications to iodinated contrast including renal insufficiency, hypersensitivity, and hyperthyroidism
* Acute severe colonic obstruction which is likely preclude safe and successful performance of CTC
* Patient who is suspicious for colonic perforation
* Pregnancy
* Phenylketonuria (contraindication to simethicone)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Colonic bubble-related image quality | within 1 month after assessment of the other primary endpoint
  Colonic bubble-specific image quality is evaluated semi-quantitatively in terms of colonic mucosal surface obscured/covered by colonic bubbles.

SECONDARY OUTCOMES:
Overall image quality | within 3 months after enrollment of all the patients and acquisition of CT colonography in all enrolled patients
  Overall image quality according to the CT Colonography Reporting and Data System. Rate of C0, i.e. polyps 1 cm or larger cannot be excluded due to insufficient technical quality, is assessed.
diagnostic performance | within 3 months after enrollment of all the patients and acquisition of CT colonography in all enrolled patients
  diagnostic performance of CT colonography for detecting colonic adenoma or carcinoma 6 mm or greater in diameter

CONTACTS AND LOCATIONS:
Overall Officials: Seong Ho Park, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea